CLINICAL TRIAL: NCT03773614
Title: Impairing Drugs and Alcohol as Risk Factors for Traumatic Injuries - a National Study on Injury Prevention
Brief Title: Impairing Drugs and Alcohol as Risk Factors for Traumatic Injuries
Acronym: IDART
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Norwegian National Trauma Registry (Unknown); Norwegian National Advisory Unit on Trauma (Unknown); Norwegian Public Roads Administration (Unknown); Norwegian Directorate of Health (Other Government); Norwegian Ministry of Transport and Communications (Unknown); Sykehuset Innlandet HF (Other)
Responsible Party: Principal Investigator, Thomas Kristiansen, Principal Investigator, Oslo University Hospital
Other Study IDs: 2017/1363
Record Dates: First submitted 2018-06-10; First posted 2018-12-12 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Trauma Injury
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Impairing drugs and alcohol are major risk factors for traumatic injuries. Still there is to date little knowledge to what extent these factors affect the epidemiology of trauma. Detailed mapping of risk factors improve targeting and efficiency of primary injury prevention. The aim of this project is therefore to facilitate injury prevention through improved data collection and analysis on impairing drugs and alcohol as a contributing and modifiable factor in injury morbidity and mortality.

Study question: What is the toxicological profile among patients with suspected severe traumatic injury? Study design: a prospective population-based and national observational study will analyse toxicology from blood samples of all trauma admission during a 12 month study period.

ELIGIBILITY:
Inclusion Criteria:

* admission to any Norwegian Trauma Hospital (n=37) AND trauma team activation, during study period

Exclusion Criteria:

* age
* foreign citizens

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All trauma patients received by trauma team at any Norwegian trauma hospital during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Presence of alcohol in blood samples. | Blood sample are collected at time of hospital admission for each participant. There is only one sample taken from each participant. Samples are consecutively analyzed during the study period. The database is analyzed after study period is completed.
  Alcohol is reported in grams per liter. Analysis of alcohol is performed with an automated enzymatic method using alcohol dehydrogenase.
Presence of impairing illicit and medicinal drugs in blood samples. | Blood sample are collected at time of hospital admission for each participant. There is only one sample taken from each participant. Samples are consecutively analyzed during the study period.
  Impairing substances are reported as nanogram per milliliter. Analysis is performed using liquid chromatography coupled with mass spectrometry.

CONTACTS AND LOCATIONS:
Locations (1):
- OsloUH, Oslo, Norway